CLINICAL TRIAL: NCT01872013
Title: Randomized, Double-blinded, Placebo-controlled, Multiple Oral Administration of ASP7991 to Non-elderly Male Subjects
Brief Title: Multiple Oral Administration of ASP7991 to Non-elderly Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 7991-CL-1002
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy; Pharmacokinetics of ASP7991
Keywords: Plasma concentration; Urinary concentration; ASP7991
MeSH Terms: interventions — ASP7991

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- low dose ASP7991 (Experimental)
  Interventions: Drug: ASP7991
- middle dose ASP7991 (Experimental)
  Interventions: Drug: ASP7991
- high dose ASP7991 (Experimental)
  Interventions: Drug: ASP7991
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7991 — oral
  Arms: high dose ASP7991; low dose ASP7991; middle dose ASP7991
Drug: Placebo — oral
  Arms: Placebo

SUMMARY:
This study is to assess the safety, tolerability, plasma concentration and pharmacodynamics of ASP7991 after multiple oral administrations to non-elderly subjects.

DETAILED DESCRIPTION:
In each step (lowest dose, middle dose, highest dose), subjects are randomly assigned in a double blinded manner to receive either ASP7991 (n=9) or Placebo (n=3) and are administered repeatedly. Once daily, the subjects are administered ASP7991 or placebo orally 30 minutes after breakfast with 150 mL water for 7 days. After the each step the sponsor evaluates the safety in the blinded manner for deciding an escalation to the step.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, as judged by the investigator/sub investigator based on the results of physical examination obtained before study drug administration
* Body weight: ≥50.0 kg, <80.0 kg
* BMI: ≥17.6, <26.4
* Serum corrected calcium concentration: ≥9.0mg/dL, <10.4 mg/dL

Exclusion Criteria:

* Received any investigational drugs in other clinical or post-marketing studies within 120 days before screening
* Donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days before screening
* Received medication (including marketed drug) within 7 days before hospitalization, vitamin preparation including vitamin D and supplement including calcium or is scheduled to receive medication
* A deviation from normal criteria range of 12-lead ECG (QT evaluation)
* A deviation from the normal range in clinical laboratory tests
* Highly sensitive cardiac troponin T (at screening): ≥0.014 ng/mL
* History of drug allergies
* Upper gastrointestinal disease (e.g. nausea, vomiting, stomachache) within 7 days before admission
* Concurrent or previous hepatic disease (e.g., viral hepatitis, drug-induced liver injury)
* Concurrent or previous endocrine disorders (e.g., hyperthyroidism, aberration in growth hormone)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The safety of ASP7991 assessed by the incidence of adverse events, vital signs, laboratory tests, 12-lead ECGs, ECGs for QT evaluation and slit lamp examination | For 96 hours after dosing

SECONDARY OUTCOMES:
Plasma concentrations unchanged drug; AUC24h, Cmax, Ctrough, tmax, t1/2, CL/F, Vz/F | For 96 hours after dosing
Urinary concentrations unchanged drug; Aelast, Aelast%, CLR | For 96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Tokyo, Japan